CLINICAL TRIAL: NCT03459417
Title: Safety and Efficacy of Intrathecally Administered Magnesium Sulfate Added to Morphine and Local Anesthetics for Major Abdominal Cancer Surgery
Brief Title: Safety and Efficacy of Intrathecally Administered Magnesium Sulfate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECI-Assuit
Record Dates: First submitted 2018-02-21; First posted 2018-03-08 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Cancer; Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intrathecal morphine+LA (Active Comparator): patients will receive intrathecal 15 mg (3 mL) of LA (hyperbaric bupivacaine 0.5%) intrathecal with 0.5 mg preservative free morphine.
  Interventions: Procedure: intrathecal morphine+LA
- intrathecal morphine+LA+Mg sulp. 50 (Active Comparator): patients will receive intrathecal 15 mg (3 mL) of LA (hyperbaric bupivacaine 0.5%) intrathecal with 0.5 mg preservative free morphine + magnesium sulfate 50 mg.
  Interventions: Procedure: intrathecal morphine+LA+ Mg sulp. 50
- intrathecal morphine+LA+ Mg sulp.100 (Active Comparator): patients will receive intrathecal 15 mg (3 mL) of LA (hyperbaric bupivacaine 0.5%) intrathecal with 0.5 mg preservative free morphine + magnesium sulfate 100 mg.
  Interventions: Procedure: intrathecal morphine+LA+ Mg sulp. 100

INTERVENTIONS:
Procedure: intrathecal morphine+LA — Lumbar puncture will be performed in the sitting position. A 25 gauge (pencil point, Braun, Melsungen, Germany) spinal needle will be introduced into the subarachnoid space at the L3-L4 lumber level midline approach with the needle orifice cephalad. Cerebrospinal fluid will be aspirated and the ready mixture will be injected to subarachnoid space over the period of 15 s, with barbotage. patients will receive intrathecal LA 15 mg (3 mL) (hyperbaric bupivacaine 0.5%) intrathecal with 0.5 mg preservative free morphine + magnesium sulfate 100 mg.
  Arms: intrathecal morphine+LA
Procedure: intrathecal morphine+LA+ Mg sulp. 50 — Lumbar puncture will be performed in the sitting position. A 25 gauge (pencil point, Braun, Melsungen, Germany) spinal needle will be introduced into the subarachnoid space at the L3-L4 lumber level midline approach with the needle orifice cephalad. Cerebrospinal fluid will be aspirated and the ready mixture will be injected to subarachnoid space over the period of 15 s, with barbotage.patients will receive intrathecal 15 mg (3 mL) of hyperbaric bupivacaine 0.5% intrathecal +0.5 mg preservative free morphine + magnesium sulphate 50 mg.
  Arms: intrathecal morphine+LA+Mg sulp. 50
Procedure: intrathecal morphine+LA+ Mg sulp. 100 — Lumbar puncture will be performed in the sitting position. A 25 gauge (pencil point, Braun, Melsungen, Germany) spinal needle will be introduced into the subarachnoid space at the L3-L4 lumber level midline approach with the needle orifice cephalad. Cerebrospinal fluid will be aspirated and the ready mixture will be injected to subarachnoid space over the period of 15 s, with barbotage.patients will receive intrathecal 15 mg (3 mL) of hyperbaric bupivacaine 0.5% intrathecal with 0.5 mg preservative free morphine + magnesium sulphate 100 mg.
  Arms: intrathecal morphine+LA+ Mg sulp.100

SUMMARY:
Magnesium sulfate safety profile has been documented by histopathological analysis in experimental studies. magnesium sulfate added to local anesthetics decrease postoperative opioid requirements.

DETAILED DESCRIPTION:
Spinal anesthesia is commonly used for the major abdominal cancer surgery because of decreasing the risks of general anesthesia.The quality and duration of sensory and motor block and decrease post operative pain is important in the major abdominal cancer surgery and patient's content satisfaction. Opioids in high doses and other drug such as clonidine and neostigmine added to local anesthetics to this purpose, but significant side effects.

Magnesium sulfate block the N- methyle -D- aspartate (NMDA) channels in a voltage-dependent way to be improve the quality and duration of spinal block. However, the use of magnesium sulfate safety profile has been documented by histopathological analysis in experimental studies. Systemic delivery of magnesium sulfate decrease postoperative opioid requirements. In experimental studies, spinal injection of magnesium sulfate reduces the respond to painful stimulus in rats.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA physical status II or III, 21-year-old or older with major abdominal cancer surgery

Exclusion Criteria:

* significant coexisting, hepatorenal, or other end organ disease, obesity (BMI > 38 kg/m2), contraindication to regional anesthesia and sensitivity to local anesthetic drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
change pain sensation using VAS scores | at 0, 4, 8, 12, 18, 24, 36 and 48 hours post operative
  pain sensation using VAS scores with movement (0-10) 0=no pain 10=worst pain ever

SECONDARY OUTCOMES:
change in MAP | at 0, 4, 8, 12, 18, 24, 36 and 48 hours post operative
  Mean arterial pressure

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No